CLINICAL TRIAL: NCT02713984
Title: A Clinical Research of CAR T Cells Targeting HER2 Positive Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Reform CAR structure due to safety consideration
Sponsor: Zhi Yang (Other)
Responsible Party: Sponsor-Investigator, Zhi Yang, Researcher of Biotherpy Center, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMMU-BTC-005
Record Dates: First submitted 2016-03-12; First posted 2016-03-21 (Estimated); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer; Ovarian Cancer; Lung Cancer; Gastric Cancer; Colorectal Cancer; Glioma; Pancreatic Cancer
Keywords: HER2 CAR-T; safety; efficiency; refractory and relapsed cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Lung Neoplasms; Stomach Neoplasms; Colorectal Neoplasms; Glioma; Pancreatic Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HER2 positive cancers (Experimental): Patients with relapsed and refractory cancer of HER2 expression will be treated with anti-HER2 CAR-T cells
  Interventions: Biological: Anti-HER2 CAR-T

INTERVENTIONS:
Biological: Anti-HER2 CAR-T — HER-2-targeting CAR-T cells infusion in HER2 positive cancers

SUMMARY:
Chimeric antigen receptor T cells (CAR-T) therapy has not yet been fully explored in solid tumors. Human epidermal growth factor receptor-2(HER2) is widely expressed in cancers. Investigators have developed anti-HER2 CAR-modified T cells and validated the efficiency targeting HER2-positive cancer in preclinical studies. This study is aimed to confirm its adverse effects including cytokine storm response and any other adverse effects. In addition, CAR-T cells persistence, tumor elimination and disease status after treatment will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory HER2 positive cancer.
2. KPS>60.
3. Life expectancy>3 months.
4. Gender unlimited, age from 18 years to 80 years.
5. Assessable lesions with a minimum size of 10mm by CT scan or MRI.
6. Acceptable organ function

   Hematology:
   * Absolute neutrophil count greater than 800/mm^3 without the support of filgrastim.
   * White blood cell (WBC) (> 2000/mm^3).
   * Platelet count greater than 50,000/mm^3.
   * Hemoglobin greater than 9.0 g/dl.

   Chemistry:
   * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less or equal to 3 times the upper limit of normal (patients without liver metastasis) or 6 times the upper limit of normal (patients with liver metastasis).
   * Serum creatinine less or equal to 3 times the upper limit of normal
   * Total bilirubin less than or equal to 3 times the upper limit of normal.
7. No other serious diseases(autoimmune disease, immunodeficiency etc.).
8. Adequate cardiac function(LVEF≥40%).
9. No other tumors.
10. Patients volunteer to participate in the research.

Exclusion Criteria:

1. Allergic to cytokines.
2. Uncontrolled active infection.
3. Acute or chronic GVHD.
4. MODS.
5. Treated with T cell inhibitor.
6. HIV affected.
7. Other situations improper for the research.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Determine the toxicity profile of the HER2 targeted CAR T cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0. | 3 years
  Observe and handle the toxicity profile of the HER2 targeted CAR T cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Survival time of Anti-HER2 CAR T cells in vivo. | 1 year
  Detect the existence of CAR-T cells in the blood of participants through qPCR or flow cytometry.
Efficacy of anti-HER2 CAR T cells to confirm the ability of CAR T cells to eliminate HER2 positive cancer cells | 12 weeks
  Evaluate the anti-tumor efficacy of CAR-T therapy by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 and Immune-Related Response Criteria（iRECIST）.
Maximum tolerated dose (MTD) of HER2 targeted CAR T cells | 4 weeks
  Determine the maximum tolerated dose of each participant through the grades of side effects.

CONTACTS AND LOCATIONS:
Overall Officials: Cheng Qian, MD,PhD, Principal Investigator — Southwest Hospital, China
Locations (1):
- Southwest Hospital of Third Millitary Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided